CLINICAL TRIAL: NCT05671367
Title: Evaluation of the Correlation Between Coronary Microvascular Resistance Based on Quantitative Flow Ratio and Major Adverse Cardiovascular Events in Patients With Obstructive Hypertrophic Cardiomyopathy: A Retrospective Cohort Study
Brief Title: Association Between Microvascular Resistance and Outcomes in Patients With Obstructive Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lihong Ma, Director of Department of Traditional Chinese Medicine, Principal Investigator, Clinical Professor, China National Center for Cardiovascular Diseases
Other Study IDs: 2022-1872
Record Dates: First submitted 2022-12-31; First posted 2023-01-04 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Microvascular Dysfunction; Hypertrophic Obstructive Cardiomyopathy; Microcirculation Resistance
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Artery without microcirculation resistance: The angiographic microvascular resistance (AMR) index was analyzed by interventional laboratory platform image analysis software (AngioPlus 2.0). AMR<2.5 mmHg*s/cm is defined as no microvascular resistance.
- Single artery with microcirculation resistance: The angiographic microvascular resistance (AMR) index was analyzed by interventional laboratory platform image analysis software (AngioPlus 2.0). AMR≥2.5 mmHg*s/cm is defined as microvascular resistance. There is only one of three major coronary arteries in 3 that meets this condition.
- Multiple arteries with microcirculation resistance: The angiographic microvascular resistance (AMR) index was analyzed by interventional laboratory platform image analysis software (AngioPlus 2.0). AMR≥2.5 mmHg*s/cm is defined as microvascular resistance. Two of the three major coronary arteries meet this condition.
- Three arteries with microcirculation resistance: The angiographic microvascular resistance (AMR) index was analyzed by interventional laboratory platform image analysis software (AngioPlus 2.0). AMR≥2.5 mmHg*s/cm is defined as microvascular resistance. All three major coronary arteries meet this condition.
- Significant microcirculation resistance: The angiographic microvascular resistance (AMR) index was analyzed by interventional laboratory platform image analysis software (AngioPlus 2.0). AMR≥2.5 mmHg*s/cm is defined as microvascular resistance. The sum of AMR of the three main arteries is greater than 7.5mmHg*s/cm

SUMMARY:
About 60% of patients with hypertrophic cardiomyopathy have microvascular dysfunction. Microvascular dysfunction is directly related to prognosis in hypertrophic cardiomyopathy. This new measurement method is microcirculation resistance (MR) based on quantitative flow ratio (QFR), which does not need a pressure guide wire on the basis of angiography. The QFR system is used to evaluate the blood vessels distal pressure and blood flow, and their ratio is microcirculation resistance (MR). The quantitative blood flow fraction measurement system was analyzed by interventional laboratory platform image analysis software (AngioPlus 2.0). This study is a single-center retrospective cohort study. Participants were selected from patients who were diagnosed with hypertrophic obstructive cardiomyopathy in Fuwai Hospital from January 2020 to November 2021. The risk factor is whether there is microcirculation resistance disorder. The outcome was the major adverse cardiovascular events related to HCM (including all-cause death, heart transplantation, left ventricular pacemaker, and heart failure readmission) that were followed up one year after angiography. Aim To further clarify whether there is a certain correlation between microvascular resistance and adverse cardiovascular prognosis.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18-80 years old;
2. Patients with hypertrophic obstructive cardiomyopathy undergoing coronary angiography. Diagnosis criteria that meet the diagnostic guidelines for hypertrophic obstructive cardiomyopathy: It usually refers to the thickness of the ventricular septum or left ventricular wall measured by two-dimensional echocardiography > 15 mm, or the thickness of > 13mm in patients with a clear family history, usually without enlargement of the left ventricular cavity, and the thickening of the left ventricular wall caused by increased loads, such as hypertension, aortic stenosis, and congenital subvalvular septum should be excluded; LVOTG>30 mmHg under quiet or exercise conditions.
3. The informed consent form for the use of sample data of patients admitted to the hospital has been signed;

Exclusion criteria:

1. No contrast examination is performed for various reasons;
2. Missing baseline important information indicators;
3. Loss of follow-up;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2017 to November 2021, patients with hypertrophic obstructive cardiomyopathy underwent coronary angiography in Fuwai Hospital.
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
The Major Adverse Cardiovascular Events related to HoCM | One-year followed up after angiography
  including all-cause death, heart transplantation, left ventricular pacemaker, heart failure readmission

SECONDARY OUTCOMES:
Scale of KCCQ-12 | One-year followed up after angiography
  KCCQ-12, a questionnaire of cardiomyopathy in Kansas City, which comes from the telephone follow-up or reexamination of cardiac rehabilitation records of departments, consists of 8 questions and 12 items, which are simplified from KCCQ-23. The score ranged from 0 to 100 points, with a higher score and better health.
Borg Index after 6MWT | One-year followed up after angiography
  Borg index reflects the dyspnea and fatigue level after 6MWT, with a standard score of 0-10. The score ranged from 0 to 10 points, and a higher score indicated a better prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lihong Ma, MD, Principal Investigator — Fuwai Hospital, China National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Authors/Task Force members; Elliott PM, Anastasakis A, Borger MA, Borggrefe M, Cecchi F, Charron P, Hagege AA, Lafont A, Limongelli G, Mahrholdt H, McKenna WJ, Mogensen J, Nihoyannopoulos P, Nistri S, Pieper PG, Pieske B, Rapezzi C, Rutten FH, Tillmanns C, Watkins H. 2014 ESC Guidelines on diagnosis and management of hypertrophic cardiomyopathy: the Task Force for the Diagnosis and Management of Hypertrophic Cardiomyopathy of the European Society of Cardiology (ESC). Eur Heart J. 2014 Oct 14;35(39):2733-79. doi: 10.1093/eurheartj/ehu284. Epub 2014 Aug 29. No abstract available. PMID 25173338
- [Background] Maron BJ, Maron MS. Hypertrophic cardiomyopathy. Lancet. 2013 Jan 19;381(9862):242-55. doi: 10.1016/S0140-6736(12)60397-3. Epub 2012 Aug 6. PMID 22874472
- [Background] Stahli BE, Erbay A, Steiner J, Klotsche J, Mochmann HC, Skurk C, Lauten A, Landmesser U, Leistner DM. Comparison of resting distal to aortic coronary pressure with angiography-based quantitative flow ratio. Int J Cardiol. 2019 Mar 15;279:12-17. doi: 10.1016/j.ijcard.2018.11.093. Epub 2018 Nov 17. PMID 30545620
- [Background] Park J, Lee JM, Koo BK, Shin ES, Nam CW, Doh JH, Hwang D, Zhang J, Hu X, Wang J, Ye F, Chen S, Yang J, Chen J, Tanaka N, Yokoi H, Matsuo H, Takashima H, Shiono Y, Akasaka T. Clinical Relevance of Functionally Insignificant Moderate Coronary Artery Stenosis Assessed by 3-Vessel Fractional Flow Reserve Measurement. J Am Heart Assoc. 2018 Feb 15;7(4):e008055. doi: 10.1161/JAHA.117.008055. PMID 29449274
- [Background] Fan Y, Fezzi S, Sun P, Ding N, Li X, Hu X, Wang S, Wijns W, Lu Z, Tu S. In Vivo Validation of a Novel Computational Approach to Assess Microcirculatory Resistance Based on a Single Angiographic View. J Pers Med. 2022 Oct 31;12(11):1798. doi: 10.3390/jpm12111798. PMID 36573725